CLINICAL TRIAL: NCT03297983
Title: Phase I, Open-label, Randomized, Two Part, Three-Period, Two-Sequence, Cross-over Study to Investigate the Relative Bioavailability of a Tablet Formulation Compared to Powder-in-Capsule of M7583 Including a Food Effect Evaluation for the Tablet in Healthy Volunteers
Brief Title: M7583 Relative Bioavailability of Tablet Compared to Powder-in-capsule
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MS200662-0017; 2017-001674-41 (EudraCT Number)
Record Dates: First submitted 2017-09-27; First posted 2017-09-29 (Actual); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Healthy
Keywords: M7583; Healthy Subjects; Cross-over

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First M7583 Tablet:Fasted, Then PiC:Fasted, Then Tablet:Fed (Experimental)
  Interventions: Drug: M7583
- First M7583 PiC:Fasted, Then Tablet:Fasted, Then Tablet:Fed (Experimental)
  Interventions: Drug: M7583

INTERVENTIONS:
Drug: M7583 — Subject will receive either M7583 PiC or M7583 tablet formulation orally under fasted conditions in part 1 followed by M7583 tablet formulation under fed condition in part 2 of the study.

SUMMARY:
This is a Phase I study consisting of 2 parts: Part 1 aims to investigate the relative bioavailability of tablet formulation (test treatment) and Powder in capsule (PiC) formulation (reference treatment) of M7583 under fasted conditions. The aim of Part 2 is to determine and compare the single dose Pharmacokinetic (PK) profile of M7583 tablet under fasted and fed conditions to assess the food effect.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females between 18 and 55 years of age (inclusive) with total body weight between 50.0 and 100.0 kilogram (kg) (inclusive) and body mass index (BMI) between 19.0 and 30.0 kilogram per meter square (kg/m2) (inclusive) at the time of the Screening examination.
* A female participant is eligible to participate if she is not pregnant, not breastfeeding.
* Females must have a negative serum pregnancy test at Screening visit and at Day -1 before randomization/first dosing.
* Men must agree to use a barrier method (specifically, male condom with or without spermicide) and to have their female partners use a highly effective method of contraception during the treatment period, and for at least 3 months after the last IMP administration. Men must also refrain from donating sperm during this period.
* Healthy as assessed by the Investigator with no clinically significant abnormality identified on physical examination or laboratory evaluation and no active clinically significant disorder, condition, infection or disease that would pose a risk to subject safety or interfere with the trial evaluation, procedures, or completion.
* Stable non-smokers for at least 3 months preceding Screening.
* Must agree not to consume any alcohol during the treatment period of the trial.
* Able and willing to give written informed consent and has signed the appropriate written informed consent form, approved by the Investigator's Independent Ethics Committee (IEC), prior to the performance of any trial activities.

Exclusion Criteria:

* History of clinically relevant disease of any organ system, that may interfere with the objectives of the trial or provide a risk to the health of the subject.
* History of chronic or recurrent acute infection or any bacterial, viral, parasitic or fungal infections within 30 days prior to Screening and at any time between Screening and admission, or hospitalization due to infection within 6 months prior to Screening.
* History of Herpes zoster within 12 months prior to Screening
* History of drug hypersensitivity, ascertained or presumptive allergy/hypersensitivity to the active drug substance and/or formulation ingredients; history of serious allergic reactions leading to hospitalization or any other hypersensitivity reaction in general, which may affect the safety of the subject and/or outcome of the trial per the Investigator's discretion.
* History of alcoholism or drug abuse within 2 years prior to Screening and the subject is unwilling to abstain from alcohol and drug of abuse during the trial
* Consumption of an average weekly intake of greater than (>) 14 drinks/week for males or > 7 drinks/week for females. One drink is equivalent to (12 g alcohol) = 5 ounces (150 milliliter (mL)) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of 40 Vol% distilled spirits.
* Positive for drugs of abuse, nicotine/cotinine or alcohol at Screening or at admission.
* Supine systolic blood pressure > 140 mmHg or less than (<) 90 mmHg, diastolic blood pressure > 90 mmHg or <50 and pulse rate >100 or ≤ 50 bpm, at admission.
* 12-Lead ECG showing a QTcF > 450 ms, PQ > 200ms, or QRS > 120 ms or other clinically relevant abnormal findings

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2017-12-06 (Actual); Study Completion 2017-12-06 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Concnetration (AUC0-t) of M7583 | pre-dose, 0.25, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 12.0, 16.0, 24.0, and 36.0 hours post-dose on Day 1 in each period
Area Under the Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUC0-∞) of M7583 | pre-dose, 0.25, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 12.0, 16.0, 24.0, and 36.0 hours post-dose on Day 1 in each period
Maximum Observed Drug Concentration (Cmax) of M7583 | pre-dose, 0.25, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 12.0, 16.0, 24.0, and 36.0 hours post-dose on Day 1 in each period

SECONDARY OUTCOMES:
Occurrence of Treatment Emergent Adverse Events (TEAEs) and Serious TEAEs | Up to Week 6
Occurrence of Subjects With TEAEs by Severity According to Qualitative Toxicity Scale Selected From National Cancer Institute - Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 | Up to Week 6
Number of Subjects with Clinically Significant Change From Baseline in Laboratory Tests, Vital Sign and 12-lead Electrocardiogram (ECG) Findings | Up to Week 6
Time to Reach the Maximum Plasma Concentration (tmax) of M7583 | pre-dose, 0.25, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 12.0, 16.0, 24.0, and 36.0 hours post-dose on Day 1 in each period
Terminal Rate Constant (λz) of M7583 | pre-dose, 0.25, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 12.0, 16.0, 24.0, and 36.0 hours post-dose on Day 1 in each period
Apparent Terminal Half-life (t1/2) of M7583 | pre-dose, 0.25, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 12.0, 16.0, 24.0, and 36.0 hours post-dose on Day 1 in each period
Total Body Clearance of Drug From Plasma Following Oral Administration (CL/f) of M7583 | pre-dose, 0.25, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 12.0, 16.0, 24.0, and 36.0 hours post-dose on Day 1 in each period
Apparent Volume of Distribution (Vz/f) of M7583 | pre-dose, 0.25, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 12.0, 16.0, 24.0, and 36.0 hours post-dose on Day 1 in each period
Area Under the M7583 Plasma Concentration-time Curve From Time Zero to 24 hours After Dosing (AUC0-24h) | pre-dose, 0.25, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 12.0, 16.0, 24.0, and 36.0 hours post-dose on Day 1 in each period
Percentage of AUC0-∞ Obtained by Extrapolation (%AUCextra) of M7583 | pre-dose, 0.25, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 12.0, 16.0, 24.0, and 36.0 hours post-dose on Day 1 in each period
Relative Bioavailability of M7583 Tablet versus M7583 PIC (Frel,T/P) | pre-dose, 0.25, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 12.0, 16.0, 24.0, and 36.0 hours post-dose on Day 1 in each period
Relative Bioavailability of M7583 Tablet Administered 30 Minutes After a Standard Breakfast Versus Tablet Administered After an Overnight Fast (Frel,Fed/Fasted) | pre-dose, 0.25, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 12.0, 16.0, 24.0, and 36.0 hours post-dose on Day 1 in each period

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- Nuvisan GmbH, Neu-Ulm, Bavaria, Germany